CLINICAL TRIAL: NCT05435430
Title: Post-COVID-19 Infection and Reproductive Health in Women Undergoing I.V.F. Treatment
Brief Title: COVID-19 Infection and Reproductive Health in Infertile Women
Acronym: COVINF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, GIUSEPPE GULLO, GIUSEPPE GULLO MD. Ph.D, University of Palermo
Other Study IDs: AOOR VILLA SOFIA CERVELLO
Record Dates: First submitted 2022-06-26; First posted 2022-06-28 (Actual); Last update posted 2022-06-28 (Actual); Status verified 2022-06

CONDITIONS: Infertility, Female
Keywords: SARS COV 19,IVF,OVARINA RESERVE,PREGNANCY
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- women with previously SARS-COV2 infection.: 2 group from 2 IVF CENTER with egual criteria :
  INCLUSION CRITERIA:
  * Women 24-43 years of age
  * Previous history of COVID-19 infection
  * INFERTILITY DIAGNOSIS
  ESCLUSION CRITERIA:
  * women with current symptoms of COVID-19 infection
  * Positive for HIV or the presence of active viral hepatitis
  * Previosuly ovarian cancer, removal of ovaries or gonadotoxic treatments
  Interventions: Other: PERSPECTIVE, MULTICENTRIC and observational

INTERVENTIONS:
Other: PERSPECTIVE, MULTICENTRIC and observational — we will enroll women with 25-45ys old and previously SARS-COV2 infection. first outcome to be investigate the impact of SARS-COV2 infection on female reproductive health and the main clinical-laboratory parameters (FSH, LH, AMH) relating to women with procreative research, in a path of medically procreation assisted programm and on any quantitative variations, duration and periodicity of the menstrual cycle after Covid infection compared to the pre-infection period.

SUMMARY:
An increased number of women has been infected by COVID-19 in the last 2 years SARS-CoV-2 infection could have a role in potential disturbances on hormon levels and human fertility Has not completely demonstrated COVID-19 effects on female reproductive function and further research can be undertaken.

The proposed multicenter study will be simple and rapid, and attractive for the scientific community.

DETAILED DESCRIPTION:
COVID-19 virus is classified as a respiratory disease that drastically changed our daily life and perspective (1) can be mainly transmitted via respiratory droplets, however, there are recently published reports suggested its ability to transmit via sexual intercourse, assisted reproductive technology (ART) treatments, pregnancy, and nursing. ART specialists should be precautious, carefully following the situation while contributing by sharing novel evidence to counsel our patients (2).

However, there are no comprehensive reviews to explore the association between COVID-19 and female fertility comprehensively.Its of major importance to provide in-depth research explaining the underlying mechanism of SARS-CoV-2 infection and its impact on human reproductive organs and fertility (3).

Ovarian reserve is a key determinant of female fertility. In this study we observe the potential effects of SARS-CoV-2 infection on the principal indicators of ovarian reserve function as anti-Müllerian hormone (AMH); basal follicle-stimulating hormone (FSH), basal luteinising hormone (LH) basal oestradiol (E2) antral follicle count (AFC).

Questions regarding the potential risks of sexual transmission during intercourse and/or application of ART, vertical transmission (throughout pregnancy, delivery, and breastfeeding), the health of pregnant and postpartum women, and fetal or postnatal health problems of neonates/children remain largely unanswered (4,5).

ELIGIBILITY:
Inclusion Criteria:

Women 24-43 years of age Previous history of COVID-19 infection INFERTILITY DIAGNOSIS

Exclusion Criteria:

Women with current symptoms of COVID-19 infection Positive for HIV or the presence of active viral hepatitis Previosuly ovarian cancer, removal of ovaries or gonadotoxic treatments

Ages: 25 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: mechanism of SARS-CoV-2 infection and its impact on human reproductive organs and fertility.
  Ovarian reserve is a key determinant of female fertility. In this study we observe the potential effects of SARS-CoV-2 infection on the principal indicators of ovarian reserve function as anti-Müllerian hormone (AMH); basal follicle-stimulating hormone (FSH), basal luteinising hormone (LH) basal oestradiol (E2) antral follicle count (AFC).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-09-30 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Main outcome | 18 months
  To investigate how the SARS-COV2 infection affects the female reproductive health and the main clinical-laboratory parameters (FSH, LH, AMH) relating to women with procreative research in a path of medically assisted procreation and any quantitative variations, duration and periodicity of the menstrual cycle after Covid infection.19 compared to the pre-infection period.

SECONDARY OUTCOMES:
secondary outcomes | 18 months
  Quantification of the number of good quality oocytes (MII) . Number of embryos on day 3 (Morula) or day 5 (blastocyst) of development transferred to the patients.
  Thickness of the endometrium at the time of embryo transfer (ET).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Gullo, MD.Ph.D, Principal Investigator — AOOR VILLA SOFIA CERVELLO
Locations (1):
- Aoor Villa Sofia Cervello, Palermo, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reis S, Xavier MR, Coelho R, Montenegro N. Psychological impact of single and multiple courses of assisted reproductive treatments in couples: a comparative study. Eur J Obstet Gynecol Reprod Biol. 2013 Nov;171(1):61-6. doi: 10.1016/j.ejogrb.2013.07.034. Epub 2013 Aug 6. PMID 23928476
- [Background] 3. World Health Organization. Coronavirus disease 2019 (COVID-2019) situation Report-49, 2020. Available: https://www.who.int/ emergencies/diseases/novel-coronavirus-2019 [Accessed 2 Sep 2020].
- [Background] Li F, Lu H, Zhang Q, Li X, Wang T, Liu Q, Yang Q, Qiang L. Impact of COVID-19 on female fertility: a systematic review and meta-analysis protocol. BMJ Open. 2021 Feb 25;11(2):e045524. doi: 10.1136/bmjopen-2020-045524. PMID 33632754
- [Background] Li R, Yin T, Fang F, Li Q, Chen J, Wang Y, Hao Y, Wu G, Duan P, Wang Y, Cheng D, Zhou Q, Zafar MI, Xiong C, Li H, Yang J, Qiao J. Potential risks of SARS-CoV-2 infection on reproductive health. Reprod Biomed Online. 2020 Jul;41(1):89-95. doi: 10.1016/j.rbmo.2020.04.018. Epub 2020 Apr 30. PMID 32466994
- [Background] Markiewicz-Gospodarek A, Wdowiak P, Czeczelewski M, Forma A, Flieger J, Januszewski J, Radzikowska-Buchner E, Baj J. The Impact of SARS-CoV-2 Infection on Fertility and Female and Male Reproductive Systems. J Clin Med. 2021 Sep 29;10(19):4520. doi: 10.3390/jcm10194520. PMID 34640536
- [Background] D'Ippolito S, Turchiano F, Vitagliano A, Scutiero G, Lanzone A, Scambia G, Greco P. Is There a Role for SARS-CoV-2/COVID-19 on the Female Reproductive System? Front Physiol. 2022 Mar 2;13:845156. doi: 10.3389/fphys.2022.845156. eCollection 2022. PMID 35309055
- [Result] Maroufizadeh S, Karimi E, Vesali S, Omani Samani R. Anxiety and depression after failure of assisted reproductive treatment among patients experiencing infertility. Int J Gynaecol Obstet. 2015 Sep;130(3):253-6. doi: 10.1016/j.ijgo.2015.03.044. Epub 2015 Jun 10. PMID 26100348